CLINICAL TRIAL: NCT00914485
Title: Using Multimedia Patient Feedback to Reduce Disparities in VA Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-194
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Provider Communication Skills Training (Other): Provider clinical communication training intervention
  Interventions: Behavioral: Provider Communication Skills Training

INTERVENTIONS:
Behavioral: Provider Communication Skills Training — Consists of 4 separate 1-hour sessions, 1 per "best act," in which physicians view 3 video-recorded performances of each act performed by trained actors of varied race/ethnicity.

SUMMARY:
The proposed research will provide important insight into two serious problems for veterans' healthcare: 1) mixed effectiveness of communication improvement interventions in the VA to date, and 2) persistence of racial/ethnic disparities in VA healthcare.

DETAILED DESCRIPTION:
The proposed research will provide important insight into two serious problems for veterans' healthcare: 1) mixed effectiveness of communication improvement interventions in the VA to date, and 2) persistence of racial/ethnic disparities in VA healthcare. We have identified 4 "best acts" of physician communication that patients believe to be most important in a clinical interaction. We propose to develop and evaluate a physician communication intervention that focuses specifically on these acts. In addition, our abundance of pilot study data from patients of various races/ethnicities enables us to create an intervention applicable to communication that spans patient race/ethnicity. Evaluating this intervention with physicians and patients in 2 independent VA primary care settings will help determine whether a patient-driven communication focus that incorporates input from patients of varied race/ethnicity can help "close the gap" in health outcomes between white and minority veterans.

We aim to (1) demonstrate the efficacy of using "best acts" of physician communication as content for an intervention to improve physician communication skills overall and reduce variation in communication with white versus racial/ethnic minority patients, and (2) assess the impact of patient experiences of "best acts" on patients' perceptual and behavioral outcomes.

We have collected data from over 200 primary care patients as they viewed a video of themselves and their physician interacting during a clinic visit. From these data, we are developing an educational intervention for physicians that focuses specifically on the 4 "best acts" we have identified. Scripts of the 4 "best acts" will be developed, and standardized patients at Baylor College of Medicine will perform the acts, which will be video recorded. We will then conduct a 2-site longitudinal observational study of 16 primary care physicians (8 at each site) and 36 patients of each physician. At the first site at 3-month intervals, physicians will attend an instruction session consisting of viewing a video of one best act and participating in group discussion, role-playing re-enactment of the act, and formulation of bulleted "take-away" points to facilitate subsequent recall. Once completed, the sequence of sessions will occur at the second site. At both sites, clinical interactions of participating physicians and patients will be audio recorded, and audio recordings will be analyzed for frequency of occurrence of the 4 "best acts." After each study visit, each patient will complete validated surveys measuring patients' perceptions of their physician on 4 affective dimensions known to impact patients' subsequent perceptual and behavioral outcomes. Efficacy will be assessed across patient demographics.

ELIGIBILITY:
Inclusion Criteria:

Any patient included in the regular panel of a participating physician at either study site who is a returning patient for that physician. Since 2 of the patient perceptual measures included require the pre-existence of a relationship with a specific physician, we will only enroll patients who have been seen by their physician before.

Exclusion Criteria:

* Physical disabilities that prohibit unassisted participation in research protocol:

  * legal blindness
  * dementia
  * severe post-traumatic stress disorder
  * schizophrenic disorder
  * Alzheimer's disease
  * bipolar disorder
  * and severe anxiety and/or mood disorders (must be documented in patient's medical record or attested to by patient, physician or charge nurse).
* Also, no patients new to VA primary care or to a given participating physician will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Adam Kelly, PhD MBA BS, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (2):
- United States (2):
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Provider Communication Skills Training
Started | 369
Completed | 369
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients participating in study from baseline through post-intervention.
Arm/Group | Provider Communication Skills Training
Number analyzed (Participants) | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 255
  >=65 years | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 338
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 207
  White | 129
  Hispanic/Latino | 30
  Other Race/Ethnicity | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Provider Use of Best Acts From Baseline to Post-Intervention
Description: Mean per-patient use of "best acts" learned during provider communication skills intervention, post-intervention minus baseline.
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: best acts per patient
Groups:
- Arm 1: Provider clinical communication training intervention
  Provider Communication Skills Training: Consists of 4 separate 1-hour sessions, 1 per "best act," in which physicians view 3 video-recorded performances of each act performed by trained actors of varied race/ethnicity.
Arm/Group | Arm 1
Number analyzed (Participants) | 369
best acts per patient | 0.3 (0.7)
Statistical Analysis 1: Comparison: Arm 1; Increase in mean, post-intervention versus baseline, across 18 providers and 369 patients; Test type: Superiority or Other; p = .03, t-test, 1 sided

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Arm/Group | Provider Communication Skills Training
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes